CLINICAL TRIAL: NCT03515798
Title: A Prospective Multicenter Open-label, Randomized Phase II Study of Pembrolizumab in Combination With Neoadjuvant EC-Paclitaxel Regimen in HER2-negative Inflammatory Breast Cancer.
Brief Title: Study of Immunotherapy in Combination With Chemotherapy in HER2-negative Inflammatory Breast Cancer
Acronym: PELICAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: MSD France (Industry); Oncodistinct (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PELICAN-IPC 2015-016; 2016-001868-11 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-05-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Inflammatory Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — pembrolizumab; Epirubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab (Experimental): EC Paclitaxel + Pembrolizumab Injection
  Interventions: Drug: Pembrolizumab Injection; Drug: neoadjuvant EC-paclitaxel chemotherapy
- Standard neoadjuvant chemotherapy (Active Comparator): EC Paclitaxel alone
  Interventions: Drug: neoadjuvant EC-paclitaxel chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab Injection — Patients will receive intravenously 1 dose of Pembrolizumab every 3 weeks
  Other Names: MK3475
  Arms: Pembrolizumab
Drug: neoadjuvant EC-paclitaxel chemotherapy — The cytotoxic regimen is a combination of dose-dense EC, followed by weekly paclitaxel
  Other Names: Epirubicine, Cyclophosphamide, Paclitaxel

SUMMARY:
This phase II multicentre randomized open-label study will assess the safety and efficacy of Pembrolizumab in combination with standard chemotherapy in inflammatory breast cancer. Pembrolizumab will be administered every 3 weeks during the neoadjuvant chemotherapy. Tissue and blood samples will be collected pre- and post-treatment for translational research.

DETAILED DESCRIPTION:
Inflammatory breast cancer (IBC) is a rare and highly aggressive subtype of locally advanced breast cancer representing approximately 5% of all breast cancers that requires immediate aggressive treatment. Significant progress has been made in recent years using a combination of treatments, including neoadjuvant chemotherapy, surgery and radiation therapy.

Accumulating data indicate a prognostic and/or predictive impact for immune-response variables in BC. Recent data, suggest that PD-L1 is overexpressed in a significant number of BC, notably in IBC and may have significant prognostic or predictive value. Furthermore it may be targeted to restore or boost functional antitumor immunity. Pembrolizumab, a PD-1-directed monoclonal antibody is already registered and has an out-standing activity in advanced melanoma and NSCLC patients, with promising results in several other tumor types, including triple-negative BC, and a favorable profile of tolerance.

Thus, potential benefits of pembrolizumab in combination with a conventional cytotoxic backbone may be considered as high in HER2-negative IBC.

The aim of the study is to assess the pathological complete response rate following neoadjuvant EC-paclitaxel chemotherapy plus pembrolizumab and to assess if neoadjuvant chemotherapy with anthracycline-based induction in combination with pembrolizumab exposes IBC patients to significant toxicity. rates.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 Evaluation of ECOG is to be performed within 7 days prior to the date of randomization. Note: may consider ECOG PS 2 if good rationale provided and discussed with Sponsor team.
3. Able to comply with the protocol,
4. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen, or any other regimen of social security
5. Patient (or legally acceptable representative if applicable) has provided written informed consent for the trial,
6. Previously untreated, histologically confirmed diagnosis of breast cancer and confirmed inflammatory breast cancer defined as follows:

   - T4d any N following American Joint Committee on Cancer (AJCC)-8th version classification: breast erythema, edema and/or peau d'orange, occupying at least 1/3 of the breast, with or without underlying palpable mass, duration of history of no more than 6 months.
7. HER2 negative tumors by immunohistochemistry (IHC 0 or 1+) or fluorescent/chromogenic in situ hybridization (FISH- or CISH-)
8. Hormone receptors status known,
9. No metastases,
10. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study treatment.
11. Adequate hematologic function: absolute neutrophil count ≥ 1.5 x 109/L AND platelets ≥ 100 x 109 AND Hb ≥ 9.0 g/dL or ≥5.6 mmol/L, Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
12. Adequate liver function: total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AND - ASAT ≤ 2.5 ULN AND ALAT ≤ 2.5 ULN,
13. Adequate kidney function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 30 mL/min for participant with creatinine levels >1.5 × institutional ULN, Creatinine clearance (CrCl) should be calculated per institutional standard.
14. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 ULN unless subject is receiving anticoagulant therapy, as long as PT or TCA is within therapeutic range of intended use of the anticoagulants,
15. Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% (isotopic or ultrasound methods),
16. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 12 months after the last dose of cyclophosphamide and 4 months after the last dose of pembrolizumab, whichever come last.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the subject
17. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period (corresponding to time needed to eliminate any study treatments plus an additional 120 days (a spermatogenesis cycle) for study treatments with risk of genotoxicity at any dose).

Exclusion Criteria:

1. Has metastatic breast cancer,
2. Has HER2-positive breast cancer,
3. Has bilateral breast cancer
4. Prior allogeneic stem cell or solid organ transplantation
5. A WOCBP who has a positive serum pregnancy test within 72 hours prior to randomiza-tion
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment, Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
7. Has known active CNS disease or carcinomatous meningitis.
8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug,
9. Has a known history of active TB (Bacillus Tuberculosis),
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients,
11. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy,
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment,
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis,
15. Has an active infection requiring systemic therapy.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator,
17. Has known psychiatric or substance abuse disorders that would interfere with coopera-tion with the requirements of the trial,
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment,
19. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).,
20. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies),
21. Has known history of Hepatitis B (e.g., HBsAg reactive) or known active Hepatitis C virus infection (e.g., HCV RNA [qualitative] is detected)
22. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Central evaluation of pathological complete response rate | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of NAST (i.e., ypT0/is, ypN0 in the current AJCC staging system)
Dose Limiting Toxicity (DLT) rates | during 21 days following the first administration of pembrolizumab
  incidence of DLT during the 21 days following the first administration of pembrolizumab in combination with EC, will be assessed separately in the first 3 patients of each stratum (HR+ and HR-). DLTs will be defined according to CTCAE.

SECONDARY OUTCOMES:
occurrence of serious adverse events and adverse events starting grade 2 or grade 1 (run-in period) | during 21 days following the first administration of pembrolizumab
  according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Local evaluation of pathological complete response rate | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  defined as absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of NAST (i.e., ypT0/is, ypN0 in the current AJCC staging system)
Invasive disease-free survival (IDFS) | 3 years
  time from surgery to the first documented occurrence of an event, defined as: Ipsilateral invasive breast tumor recurrence, Ipsilateral local-regional invasive breast cancer recurrence, Distant recurrence, Contralateral invasive breast cancer, Death from any cause
Invasive disease-free survival (IDFS) | 5 years
  time from surgery to the first documented occurrence of an event, defined as: Ipsilateral invasive breast tumor recurrence, Ipsilateral local-regional invasive breast cancer recurrence, Distant recurrence, Contralateral invasive breast cancer, Death from any cause
Event free survival (EFS) | 3 years
  time from randomization to disease progression, disease recurrence (local, regional, distant, or contralateral [invasive or non invasive]), or death from any cause)
Event free survival (EFS) | 5 years
  time from randomization to disease progression, disease recurrence (local, regional, distant, or contralateral [invasive or non invasive]), or death from any cause)
Overall survival (OS) | 3 years
  time from randomization to death from any cause
Overall survival (OS) | 5 years
  time from randomization to death from any cause

OTHER OUTCOMES:
Evaluation of PD-L1 expression in pre, per and post-treatment tissue | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  by IHC and mass spectrometry-based proteomics; and in plasma samples using quantitative proteomics,
Measurement of baseline Circulating tumor cells for prospective validation of their prognostic value in IBC | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  Measurement of baseline CTC for prospective validation of their prognostic value in IBC
Disease monitoring | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  Purification of ctDNA and specific sequencing for disease monitoring.
Identification of mechanisms of treatment resistance | Following completion of neoadjuvant systemic treatment, an average of 24 weeks
  Immune profiling, NGS and mouse xenografing for ex-vivo phenotypic approaches on post-treatment residual disease in order to identify mechanisms of resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Goncalves, Pr, Principal Investigator — Institut Paoli-Calmettes
Locations (12):
- France (12):
  - Clinique de L'Europe, Amiens
  - Institut Sainte Catherine, Avignon
  - Institut BERGONIE, Bordeaux
  - CENTRE Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Institut Curie hopital rene huguenin, Saint-Cloud
  - Institut de cancérologie de la loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - IUCT-Oncopole Institut Claudius Rigaud, Toulouse

REFERENCES:
- [Background] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Background] Binder-Foucard F, Rasamimanana Cerf N, Belot A, Bossard N. Estimation nationale de l'incidence et de la mortalité par cancer en France entre 1980 et 2012. Étude à partir des registres des cancers du réseau Francim. Partie 1 - Tumeurs solides-Synthèse. In: http://www.invs.sante.fr. 2013.
- [Background] Chang S, Parker SL, Pham T, Buzdar AU, Hursting SD. Inflammatory breast carcinoma incidence and survival: the surveillance, epidemiology, and end results program of the National Cancer Institute, 1975-1992. Cancer. 1998 Jun 15;82(12):2366-72. PMID 9635529
- [Background] Dawood S, Merajver SD, Viens P, Vermeulen PB, Swain SM, Buchholz TA, Dirix LY, Levine PH, Lucci A, Krishnamurthy S, Robertson FM, Woodward WA, Yang WT, Ueno NT, Cristofanilli M. International expert panel on inflammatory breast cancer: consensus statement for standardized diagnosis and treatment. Ann Oncol. 2011 Mar;22(3):515-523. doi: 10.1093/annonc/mdq345. Epub 2010 Jul 5. PMID 20603440
- [Background] Cristofanilli M, Valero V, Buzdar AU, Kau SW, Broglio KR, Gonzalez-Angulo AM, Sneige N, Islam R, Ueno NT, Buchholz TA, Singletary SE, Hortobagyi GN. Inflammatory breast cancer (IBC) and patterns of recurrence: understanding the biology of a unique disease. Cancer. 2007 Oct 1;110(7):1436-44. doi: 10.1002/cncr.22927. PMID 17694554
- [Background] McCarthy NJ, Yang X, Linnoila IR, Merino MJ, Hewitt SM, Parr AL, Paik S, Steinberg SM, Hartmann DP, Mourali N, Levine PH, Swain SM. Microvessel density, expression of estrogen receptor alpha, MIB-1, p53, and c-erbB-2 in inflammatory breast cancer. Clin Cancer Res. 2002 Dec;8(12):3857-62. PMID 12473600
- [Background] Lerebours F, Bieche I, Lidereau R. Update on inflammatory breast cancer. Breast Cancer Res. 2005;7(2):52-8. doi: 10.1186/bcr997. Epub 2005 Jan 20. PMID 15743511
- [Background] Chevallier B, Bastit P, Graic Y, Menard JF, Dauce JP, Julien JP, Clavier B, Kunlin A, D'Anjou J. The Centre H. Becquerel studies in inflammatory non metastatic breast cancer. Combined modality approach in 178 patients. Br J Cancer. 1993 Mar;67(3):594-601. doi: 10.1038/bjc.1993.109. PMID 8439510
- [Background] Rouesse J, Friedman S, Sarrazin D, Mouriesse H, Le Chevalier T, Arriagada R, Spielmann M, Papacharalambous A, May-Levin F. Primary chemotherapy in the treatment of inflammatory breast carcinoma: a study of 230 cases from the Institut Gustave-Roussy. J Clin Oncol. 1986 Dec;4(12):1765-71. doi: 10.1200/JCO.1986.4.12.1765. PMID 3783202
- [Background] Brun B, Otmezguine Y, Feuilhade F, Julien M, Lebourgeois JP, Calitchi E, Roucayrol AM, Ganem G, Huart J, Pierquin B. Treatment of inflammatory breast cancer with combination chemotherapy and mastectomy versus breast conservation. Cancer. 1988 Mar 15;61(6):1096-103. doi: 10.1002/1097-0142(19880315)61:63.0.co;2-y. PMID 3342369
- [Background] Jaiyesimi IA, Buzdar AU, Hortobagyi G. Inflammatory breast cancer: a review. J Clin Oncol. 1992 Jun;10(6):1014-24. doi: 10.1200/JCO.1992.10.6.1014. PMID 1588366
- [Background] Cristofanilli M, Buzdar AU, Sneige N, Smith T, Wasaff B, Ibrahim N, Booser D, Rivera E, Murray JL, Valero V, Ueno N, Singletary ES, Hunt K, Strom E, McNeese M, Stelling C, Hortobagyi GN. Paclitaxel in the multimodality treatment for inflammatory breast carcinoma. Cancer. 2001 Oct 1;92(7):1775-82. doi: 10.1002/1097-0142(20011001)92:73.0.co;2-e. PMID 11745249
- [Background] Cristofanilli M, Gonzalez-Angulo AM, Buzdar AU, Kau SW, Frye DK, Hortobagyi GN. Paclitaxel improves the prognosis in estrogen receptor negative inflammatory breast cancer: the M. D. Anderson Cancer Center experience. Clin Breast Cancer. 2004 Feb;4(6):415-9. doi: 10.3816/cbc.2004.n.004. PMID 15023242
- [Background] de Matteis A, Nuzzo F, D'Aiuto G, Labonia V, Landi G, Rossi E, Mastro AA, Botti G, De Maio E, Perrone F. Docetaxel plus epidoxorubicin as neoadjuvant treatment in patients with large operable or locally advanced carcinoma of the breast: a single-center, phase II study. Cancer. 2002 Feb 15;94(4):895-901. doi: 10.1002/cncr.20335.abs. PMID 11920456
- [Background] Gradishar WJ, Wedam SB, Jahanzeb M, Erban J, Limentani SA, Tsai KT, Olsen SR, Swain SM. Neoadjuvant docetaxel followed by adjuvant doxorubicin and cyclophosphamide in patients with stage III breast cancer. Ann Oncol. 2005 Aug;16(8):1297-304. doi: 10.1093/annonc/mdi254. Epub 2005 May 19. PMID 15905305
- [Background] Espinosa E, Morales S, Borrega P, Casas A, Madronal C, Machengs I, Illarramendi JA, Lizon J, Moreno JA, Belon J, Janariz J, de la Puente M, Checa T, Mel JR, Gonzalez Baron M. Docetaxel and high-dose epirubicin as neoadjuvant chemotherapy in locally advanced breast cancer. Cancer Chemother Pharmacol. 2004 Dec;54(6):546-52. doi: 10.1007/s00280-004-0830-1. Epub 2004 Aug 17. PMID 15316749
- [Background] Reitsamer R, Peintinger F, Prokop E, Hitzl W. Pathological complete response rates comparing 3 versus 6 cycles of epidoxorubicin and docetaxel in the neoadjuvant setting of patients with stage II and III breast cancer. Anticancer Drugs. 2005 Sep;16(8):867-70. doi: 10.1097/01.cad.0000173475.59616.b4. PMID 16096435
- [Background] Smith IC, Heys SD, Hutcheon AW, Miller ID, Payne S, Gilbert FJ, Ah-See AK, Eremin O, Walker LG, Sarkar TK, Eggleton SP, Ogston KN. Neoadjuvant chemotherapy in breast cancer: significantly enhanced response with docetaxel. J Clin Oncol. 2002 Mar 15;20(6):1456-66. doi: 10.1200/JCO.2002.20.6.1456. PMID 11896092
- [Background] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Background] Goncalves A, Pierga JY, Ferrero JM, Mouret-Reynier MA, Bachelot T, Delva R, Fabbro M, Lerebours F, Lotz JP, Linassier C, Dohollou N, Eymard JC, Leduc B, Lemonnier J, Martin AL, Boher JM, Viens P, Roche H. UNICANCER-PEGASE 07 study: a randomized phase III trial evaluating postoperative docetaxel-5FU regimen after neoadjuvant dose-intense chemotherapy for treatment of inflammatory breast cancer. Ann Oncol. 2015 Aug;26(8):1692-7. doi: 10.1093/annonc/mdv216. Epub 2015 May 5. PMID 25943350
- [Background] Masuda H, Brewer TM, Liu DD, Iwamoto T, Shen Y, Hsu L, Willey JS, Gonzalez-Angulo AM, Chavez-MacGregor M, Fouad TM, Woodward WA, Reuben JM, Valero V, Alvarez RH, Hortobagyi GN, Ueno NT. Long-term treatment efficacy in primary inflammatory breast cancer by hormonal receptor- and HER2-defined subtypes. Ann Oncol. 2014 Feb;25(2):384-91. doi: 10.1093/annonc/mdt525. Epub 2013 Dec 18. PMID 24351399
- [Background] Gianni L, Eiermann W, Semiglazov V, Manikhas A, Lluch A, Tjulandin S, Zambetti M, Vazquez F, Byakhow M, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Baronio R, Feyereislova A, Barton C, Valagussa P, Baselga J. Neoadjuvant chemotherapy with trastuzumab followed by adjuvant trastuzumab versus neoadjuvant chemotherapy alone, in patients with HER2-positive locally advanced breast cancer (the NOAH trial): a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet. 2010 Jan 30;375(9712):377-84. doi: 10.1016/S0140-6736(09)61964-4. PMID 20113825
- [Background] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890
- [Background] Baselga J, Bradbury I, Eidtmann H, Di Cosimo S, de Azambuja E, Aura C, Gomez H, Dinh P, Fauria K, Van Dooren V, Aktan G, Goldhirsch A, Chang TW, Horvath Z, Coccia-Portugal M, Domont J, Tseng LM, Kunz G, Sohn JH, Semiglazov V, Lerzo G, Palacova M, Probachai V, Pusztai L, Untch M, Gelber RD, Piccart-Gebhart M; NeoALTTO Study Team. Lapatinib with trastuzumab for HER2-positive early breast cancer (NeoALTTO): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2012 Feb 18;379(9816):633-40. doi: 10.1016/S0140-6736(11)61847-3. Epub 2012 Jan 17. PMID 22257673
- [Background] Pierga JY, Petit T, Delozier T, Ferrero JM, Campone M, Gligorov J, Lerebours F, Roche H, Bachelot T, Charafe-Jauffret E, Pavlyuk M, Kraemer S, Bidard FC, Viens P. Neoadjuvant bevacizumab, trastuzumab, and chemotherapy for primary inflammatory HER2-positive breast cancer (BEVERLY-2): an open-label, single-arm phase 2 study. Lancet Oncol. 2012 Apr;13(4):375-84. doi: 10.1016/S1470-2045(12)70049-9. Epub 2012 Feb 28. PMID 22377126
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Mei Z, Liu Y, Liu C, Cui A, Liang Z, Wang G, Peng H, Cui L, Li C. Tumour-infiltrating inflammation and prognosis in colorectal cancer: systematic review and meta-analysis. Br J Cancer. 2014 Mar 18;110(6):1595-605. doi: 10.1038/bjc.2014.46. Epub 2014 Feb 6. PMID 24504370
- [Background] Salgado R, Denkert C, Demaria S, Sirtaine N, Klauschen F, Pruneri G, Wienert S, Van den Eynden G, Baehner FL, Penault-Llorca F, Perez EA, Thompson EA, Symmans WF, Richardson AL, Brock J, Criscitiello C, Bailey H, Ignatiadis M, Floris G, Sparano J, Kos Z, Nielsen T, Rimm DL, Allison KH, Reis-Filho JS, Loibl S, Sotiriou C, Viale G, Badve S, Adams S, Willard-Gallo K, Loi S; International TILs Working Group 2014. The evaluation of tumor-infiltrating lymphocytes (TILs) in breast cancer: recommendations by an International TILs Working Group 2014. Ann Oncol. 2015 Feb;26(2):259-71. doi: 10.1093/annonc/mdu450. Epub 2014 Sep 11. PMID 25214542
- [Background] Schatton T, Scolyer RA, Thompson JF, Mihm MC Jr. Tumor-infiltrating lymphocytes and their significance in melanoma prognosis. Methods Mol Biol. 2014;1102:287-324. doi: 10.1007/978-1-62703-727-3_16. PMID 24258985
- [Background] Gooden MJ, de Bock GH, Leffers N, Daemen T, Nijman HW. The prognostic influence of tumour-infiltrating lymphocytes in cancer: a systematic review with meta-analysis. Br J Cancer. 2011 Jun 28;105(1):93-103. doi: 10.1038/bjc.2011.189. Epub 2011 May 31. PMID 21629244
- [Background] Ahmadzadeh M, Johnson LA, Heemskerk B, Wunderlich JR, Dudley ME, White DE, Rosenberg SA. Tumor antigen-specific CD8 T cells infiltrating the tumor express high levels of PD-1 and are functionally impaired. Blood. 2009 Aug 20;114(8):1537-44. doi: 10.1182/blood-2008-12-195792. Epub 2009 May 7. PMID 19423728
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Francisco LM, Salinas VH, Brown KE, Vanguri VK, Freeman GJ, Kuchroo VK, Sharpe AH. PD-L1 regulates the development, maintenance, and function of induced regulatory T cells. J Exp Med. 2009 Dec 21;206(13):3015-29. doi: 10.1084/jem.20090847. Epub 2009 Dec 14. PMID 20008522
- [Background] Hamel KM, Cao Y, Wang Y, Rodeghero R, Kobezda T, Chen L, Finnegan A. B7-H1 expression on non-B and non-T cells promotes distinct effects on T- and B-cell responses in autoimmune arthritis. Eur J Immunol. 2010 Nov;40(11):3117-27. doi: 10.1002/eji.201040690. Epub 2010 Oct 27. PMID 21061440
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Reiss KA, Forde PM, Brahmer JR. Harnessing the power of the immune system via blockade of PD-1 and PD-L1: a promising new anticancer strategy. Immunotherapy. 2014;6(4):459-75. doi: 10.2217/imt.14.9. PMID 24815784
- [Background] Denkert C, Loibl S, Noske A, Roller M, Muller BM, Komor M, Budczies J, Darb-Esfahani S, Kronenwett R, Hanusch C, von Torne C, Weichert W, Engels K, Solbach C, Schrader I, Dietel M, von Minckwitz G. Tumor-associated lymphocytes as an independent predictor of response to neoadjuvant chemotherapy in breast cancer. J Clin Oncol. 2010 Jan 1;28(1):105-13. doi: 10.1200/JCO.2009.23.7370. Epub 2009 Nov 16. PMID 19917869
- [Background] Loi S, Michiels S, Salgado R, Sirtaine N, Jose V, Fumagalli D, Kellokumpu-Lehtinen PL, Bono P, Kataja V, Desmedt C, Piccart MJ, Loibl S, Denkert C, Smyth MJ, Joensuu H, Sotiriou C. Tumor infiltrating lymphocytes are prognostic in triple negative breast cancer and predictive for trastuzumab benefit in early breast cancer: results from the FinHER trial. Ann Oncol. 2014 Aug;25(8):1544-50. doi: 10.1093/annonc/mdu112. Epub 2014 Mar 7. PMID 24608200
- [Background] Ali HR, Provenzano E, Dawson SJ, Blows FM, Liu B, Shah M, Earl HM, Poole CJ, Hiller L, Dunn JA, Bowden SJ, Twelves C, Bartlett JM, Mahmoud SM, Rakha E, Ellis IO, Liu S, Gao D, Nielsen TO, Pharoah PD, Caldas C. Association between CD8+ T-cell infiltration and breast cancer survival in 12,439 patients. Ann Oncol. 2014 Aug;25(8):1536-43. doi: 10.1093/annonc/mdu191. Epub 2014 Jun 9. PMID 24915873
- [Background] Rody A, Holtrich U, Pusztai L, Liedtke C, Gaetje R, Ruckhaeberle E, Solbach C, Hanker L, Ahr A, Metzler D, Engels K, Karn T, Kaufmann M. T-cell metagene predicts a favorable prognosis in estrogen receptor-negative and HER2-positive breast cancers. Breast Cancer Res. 2009;11(2):R15. doi: 10.1186/bcr2234. Epub 2009 Mar 9. PMID 19272155
- [Background] Teschendorff AE, Miremadi A, Pinder SE, Ellis IO, Caldas C. An immune response gene expression module identifies a good prognosis subtype in estrogen receptor negative breast cancer. Genome Biol. 2007;8(8):R157. doi: 10.1186/gb-2007-8-8-r157. PMID 17683518
- [Background] Sabatier R, Finetti P, Mamessier E, Raynaud S, Cervera N, Lambaudie E, Jacquemier J, Viens P, Birnbaum D, Bertucci F. Kinome expression profiling and prognosis of basal breast cancers. Mol Cancer. 2011 Jul 21;10:86. doi: 10.1186/1476-4598-10-86. PMID 21777462
- [Background] Sabatier R, Finetti P, Cervera N, Lambaudie E, Esterni B, Mamessier E, Tallet A, Chabannon C, Extra JM, Jacquemier J, Viens P, Birnbaum D, Bertucci F. A gene expression signature identifies two prognostic subgroups of basal breast cancer. Breast Cancer Res Treat. 2011 Apr;126(2):407-20. doi: 10.1007/s10549-010-0897-9. Epub 2010 May 21. PMID 20490655
- [Background] Demaria S, Volm MD, Shapiro RL, Yee HT, Oratz R, Formenti SC, Muggia F, Symmans WF. Development of tumor-infiltrating lymphocytes in breast cancer after neoadjuvant paclitaxel chemotherapy. Clin Cancer Res. 2001 Oct;7(10):3025-30. PMID 11595690
- [Background] Ladoire S, Mignot G, Dabakuyo S, Arnould L, Apetoh L, Rebe C, Coudert B, Martin F, Bizollon MH, Vanoli A, Coutant C, Fumoleau P, Bonnetain F, Ghiringhelli F. In situ immune response after neoadjuvant chemotherapy for breast cancer predicts survival. J Pathol. 2011 Jul;224(3):389-400. doi: 10.1002/path.2866. Epub 2011 Mar 25. PMID 21437909
- [Background] Ghebeh H, Mohammed S, Al-Omair A, Qattan A, Lehe C, Al-Qudaihi G, Elkum N, Alshabanah M, Bin Amer S, Tulbah A, Ajarim D, Al-Tweigeri T, Dermime S. The B7-H1 (PD-L1) T lymphocyte-inhibitory molecule is expressed in breast cancer patients with infiltrating ductal carcinoma: correlation with important high-risk prognostic factors. Neoplasia. 2006 Mar;8(3):190-8. doi: 10.1593/neo.05733. PMID 16611412
- [Background] Ghebeh H, Tulbah A, Mohammed S, Elkum N, Bin Amer SM, Al-Tweigeri T, Dermime S. Expression of B7-H1 in breast cancer patients is strongly associated with high proliferative Ki-67-expressing tumor cells. Int J Cancer. 2007 Aug 15;121(4):751-8. doi: 10.1002/ijc.22703. PMID 17415709
- [Background] Ghebeh H, Barhoush E, Tulbah A, Elkum N, Al-Tweigeri T, Dermime S. FOXP3+ Tregs and B7-H1+/PD-1+ T lymphocytes co-infiltrate the tumor tissues of high-risk breast cancer patients: Implication for immunotherapy. BMC Cancer. 2008 Feb 23;8:57. doi: 10.1186/1471-2407-8-57. PMID 18294387
- [Background] Schalper KA, Velcheti V, Carvajal D, Wimberly H, Brown J, Pusztai L, Rimm DL. In situ tumor PD-L1 mRNA expression is associated with increased TILs and better outcome in breast carcinomas. Clin Cancer Res. 2014 May 15;20(10):2773-82. doi: 10.1158/1078-0432.CCR-13-2702. Epub 2014 Mar 19. PMID 24647569
- [Background] Soliman H, Khalil F, Antonia S. PD-L1 expression is increased in a subset of basal type breast cancer cells. PLoS One. 2014 Feb 14;9(2):e88557. doi: 10.1371/journal.pone.0088557. eCollection 2014. PMID 24551119
- [Background] Mittendorf EA, Philips AV, Meric-Bernstam F, Qiao N, Wu Y, Harrington S, Su X, Wang Y, Gonzalez-Angulo AM, Akcakanat A, Chawla A, Curran M, Hwu P, Sharma P, Litton JK, Molldrem JJ, Alatrash G. PD-L1 expression in triple-negative breast cancer. Cancer Immunol Res. 2014 Apr;2(4):361-70. doi: 10.1158/2326-6066.CIR-13-0127. Epub 2014 Jan 10. PMID 24764583
- [Background] Sabatier R, Finetti P, Mamessier E, Adelaide J, Chaffanet M, Ali HR, Viens P, Caldas C, Birnbaum D, Bertucci F. Prognostic and predictive value of PDL1 expression in breast cancer. Oncotarget. 2015 Mar 10;6(7):5449-64. doi: 10.18632/oncotarget.3216. PMID 25669979
- [Background] Wimberly H, Brown JR, Schalper K, Haack H, Silver MR, Nixon C, Bossuyt V, Pusztai L, Lannin DR, Rimm DL. PD-L1 Expression Correlates with Tumor-Infiltrating Lymphocytes and Response to Neoadjuvant Chemotherapy in Breast Cancer. Cancer Immunol Res. 2015 Apr;3(4):326-32. doi: 10.1158/2326-6066.CIR-14-0133. Epub 2014 Dec 19. PMID 25527356
- [Background] Bertucci F, Finetti P, Colpaert C, Mamessier E, Parizel M, Dirix L, Viens P, Birnbaum D, van Laere S. PDL1 expression in inflammatory breast cancer is frequent and predicts for the pathological response to chemotherapy. Oncotarget. 2015 May 30;6(15):13506-19. doi: 10.18632/oncotarget.3642. PMID 25940795
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, Gajewski TF. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004 Feb 1;64(3):1140-5. doi: 10.1158/0008-5472.can-03-3259. PMID 14871849
- [Background] Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer--preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010 Oct;37(5):430-9. doi: 10.1053/j.seminoncol.2010.09.005. PMID 21074057
- [Background] Strome SE, Dong H, Tamura H, Voss SG, Flies DB, Tamada K, Salomao D, Cheville J, Hirano F, Lin W, Kasperbauer JL, Ballman KV, Chen L. B7-H1 blockade augments adoptive T-cell immunotherapy for squamous cell carcinoma. Cancer Res. 2003 Oct 1;63(19):6501-5. PMID 14559843
- [Background] Spranger S, Koblish HK, Horton B, Scherle PA, Newton R, Gajewski TF. Mechanism of tumor rejection with doublets of CTLA-4, PD-1/PD-L1, or IDO blockade involves restored IL-2 production and proliferation of CD8(+) T cells directly within the tumor microenvironment. J Immunother Cancer. 2014 Feb 18;2:3. doi: 10.1186/2051-1426-2-3. eCollection 2014. PMID 24829760
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Derived] Bertucci A, Bertucci F, Zemmour C, Lerebours F, Pierga JY, Levy C, Dalenc F, Grenier J, Petit T, Berline M, Goncalves A. PELICAN-IPC 2015-016/Oncodistinct-003: A Prospective, Multicenter, Open-Label, Randomized, Non-Comparative, Phase II Study of Pembrolizumab in Combination With Neo Adjuvant EC-Paclitaxel Regimen in HER2-Negative Inflammatory Breast Cancer. Front Oncol. 2020 Nov 25;10:575978. doi: 10.3389/fonc.2020.575978. eCollection 2020. PMID 33330051
- See also: Official Website of the sponsor — http://institutpaolicalmettes.fr